CLINICAL TRIAL: NCT04516291
Title: A Phase 2b Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Dose-Ranging Study to Assess the Efficacy, Safety, and Tolerability of Vupanorsen (PF-07285557) in Statin-Treated Participants With Dyslipidemia
Brief Title: A Dose-Ranging Study With Vupanorsen (TRANSLATE-TIMI 70)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: The TIMI Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C4491011; 2020-002796-35 (EudraCT Number)
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Results first posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Dyslipidemias; Hyperlipidemias; Hyperlipoproteinemias
Keywords: Primary hyperlipidemia; Mixed dyslipidemia; Lipid Metabolism Disorders; Metabolic Diseases
MeSH Terms: conditions — Dyslipidemias; Hyperlipidemias; Hyperlipoproteinemias; Lipid Metabolism Disorders; Metabolic Diseases | interventions — vupanorsen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Placebo (Placebo Comparator): No drug
  Interventions: Drug: Placebo
- Vupanorsen 80 mg every 4 weeks (Experimental): 80 milligrams (mg) given subcutaneously every 4 weeks.
  Interventions: Drug: Vupanorsen
- Vupanorsen 60 mg every 2 weeks (Experimental): 60 mg given subcutaneously every 2 weeks.
  Interventions: Drug: Vupanorsen
- Vupanorsen 120 mg every 4 weeks (Experimental): 120 mg given subcutaneously every 4 weeks.
  Interventions: Drug: Vupanorsen
- Vupanorsen 80 mg every 2 weeks (Experimental): 80 mg given subcutaneously every 2 weeks.
  Interventions: Drug: Vupanorsen
- Vupanorsen 160 mg every 4 weeks (Experimental): 160 mg given subcutaneously every 4 weeks.
  Interventions: Drug: Vupanorsen
- Vupanorsen 120 mg every 2 weeks (Experimental): 120 mg given subcutaneously every 2 weeks.
  Interventions: Drug: Vupanorsen
- Vupanorsen 160 mg every 2 weeks (Experimental): 160 mg given subcutaneously every 2 weeks.
  Interventions: Drug: Vupanorsen

INTERVENTIONS:
Drug: Vupanorsen — Vupanorsen and placebo will be provided as prefilled syringes packaged and dispensed in cartons with tamper-evident seals. Only single-use syringes will be used.
  Other Names: PF-07285557
  Arms: Vupanorsen 120 mg every 2 weeks; Vupanorsen 120 mg every 4 weeks; Vupanorsen 160 mg every 2 weeks; Vupanorsen 160 mg every 4 weeks; Vupanorsen 60 mg every 2 weeks; Vupanorsen 80 mg every 2 weeks; Vupanorsen 80 mg every 4 weeks
Drug: Placebo — Vupanorsen and placebo will be provided as prefilled syringes packaged and dispensed in cartons with tamper-evident seals. Only single-use syringes will be used.
  Arms: Placebo

SUMMARY:
This is a multicenter, Phase 2b, double-blind, placebo-controlled, parallel group study to provide data on efficacy, safety, tolerability, and pharmacokinetics (PK) of PF-07285557 (hereafter, vupanorsen) administered subcutaneously (SC) at various doses and regimens in participants with dyslipidemia, defined in this study as participants with elevated non-HDL-C and TG who are receiving a stable dose of a statin.

This study is also known as TaRgeting ANGPTL3 with an aNtiSense oLigonucleotide in AdulTs with dyslipidEmia (TRANSLATE-TIMI 70).

DETAILED DESCRIPTION:
This study is intended to enable selection of a dose(s) for future development of vupanorsen for cardiovascular (CV) risk reduction and hypertriglyceridemia.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged ≥40 years at Screening.
2. Fasting non-HDL-C at Screening ≥100 mg/dL.
3. Fasting TG at Screening of 150 to 500 mg/dL, inclusive, which may be repeated once if deemed necessary.
4. Participants must be on a stable dose of a statin for at least 1 month before Screening and plan to remain on the same medication and dose for the duration of the study.
5. Body weight ≥50 kg and ≤136 kg at Screening.
6. Capable of giving signed informed consent.

Exclusion Criteria:

1. Participant has active liver disease (other than NAFLD or NASH, which are permitted), including chronic active hepatitis B or C or primary biliary cirrhosis.
2. Uncontrolled hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure >100 mmHg). Note: participants who are on an anti-hypertensive medication to treat hypertension should be on a stable dose at least 1 month prior to Screening. The investigator should ensure participant took anti-hypertensive medication as prescribed prior to evaluation of blood pressure.
3. Participant with a known bleeding diathesis or coagulation disorder.
4. Participants with ANY of the following abnormalities in clinical laboratory tests at Screening, as assessed by the central laboratory and confirmed by a single repeat test, if deemed necessary: HbA1c ≥9.5% eGFR <30 mL/min/1.73 m2 (as determined by the CKD-Epi equation) ALT or AST >2 × ULN Total bilirubin ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have a direct bilirubin measured and would be eligible for this study provided the direct bilirubin is ≤ULN Platelet count <LLN
5. History of clinically significant acute cardiac event within 3 months before Screening (includes ischemic stroke, transient ischemic attack, myocardial infarction, revascularization procedures, hospitalization for heart failure).
6. Presence of New York Heart Association Functional Classification IV heart failure symptoms at Screening.
7. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated.
8. Current history of alcoholism or drug addiction according to Diagnostic and Statistical Manual of Mental Disorders IV criteria within 12 months prior to Screening. Use of any recreational drugs within 12 months prior to Screening.
9. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

   Prior/Concomitant Therapy:
10. Prior treatment at any time with vupanorsen.
11. Prior treatment with any oligonucleotide (including small interfering ribonucleic acid) within 6 months of Screening or prior treatment with inclisiran within 12 months of Screening.
12. Use of TG lowering medication (eg, Vascepa [icosapent ethyl]), non-prescription dietary supplements (eg, fish oil) or other cholesterol lowering medication (eg, fibric acid derivatives, niacin, PCSK9 inhibitors, bile acid sequestrants, bempedoic acid) 30 days prior to Screening, other than statins and ezetimibe.
13. Use of warfarin or other coumarins, direct thrombin inhibitors, Factor Xa inhibitors, heparins or heparinoids 30 days prior to Screening.

    Prior/Concurrent Clinical Study Experience:
14. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).

    Diagnostic Assessments:
15. Participant has a clinically significant ECG abnormality during the Screening Period that requires further diagnostic evaluation or intervention (eg, new, clinically significant arrhythmia or a conduction disturbance).

    Other Exclusions
16. Unstable weight (>5% shift in past month) or plan to start a diet for the purpose of significant weight loss.
17. Hypersensitivity to the active substance or to any of the excipients or GalNAc.
18. Any major surgery, including bariatric surgery, within 3 months of Screening.
19. Participants with conditions contraindicated for MRI procedures including pacemakers or aneurysm clips; the presence of MRI incompatible implanted devices; metallic foreign bodies; metal tattoos (including permanent make-up); or severe claustrophobia impacting the ability to perform MRI. Participants who may require mild sedative or anxiolytic in order to complete the MRI may be enrolled.
20. Participants unwilling or unable to comply with study procedures, including follow-up, as specified by this protocol, or unwillingness to cooperate fully with the Investigator.
21. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (112):
- United States (59):
  - Horizon Clinical Research Associates, PLLC, Gilbert, Arizona
  - Scottsdale Medical Imaging Research, LLC, Gilbert, Arizona
  - CARTI, Little Rock, Arkansas
  - Atria Clinical Research, Little Rock, Arkansas
  - Clinical Trials Research, Lincoln, California
  - Diagnostic Radiological Imaging, Sacramento, California
  - West Coast Radiology, Santa Ana, California
  - University Clinical Investigators, Inc., Tustin, California
  - Tower Radiology Parsons, Brandon, Florida
  - Tower Radiology, Brandon, Florida
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Precision Imaging Centers, Jacksonville, Florida
  - Care Partners Clinical Research, LLC, Jacksonville, Florida
  - Advanced Research Institute, Inc., New Port Richey, Florida
  - Sand Lakes Imaging, Orlando, Florida
  - St Johns Center for Clinical Research, Saint Augustine, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Alliance for Multispecialty Research, LLC, El Dorado, Kansas
  - Susan B. Allen Memorial Hospital, El Dorado, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Heartland Imaging, Louisville, Kentucky
  - Maryland Cardiovascular Specialists, Baltimore, Maryland
  - Seton Imaging Center, Baltimore, Maryland
  - Lahey Clinic Hospital and Medical Center, Burlington, Massachusetts
  - Pentucket Medical Associates, Haverhill, Massachusetts
  - Regions Hospital - HealthPartners, Saint Paul, Minnesota
  - Viable Research Management LLC, Henderson, Nevada
  - Pueblo Medical Imaging, Henderson, Nevada
  - Capital Cardiology Associates, Albany, New York
  - ImageCare Latham, Latham, New York
  - Randolph Health Internal Medicine, Asheboro, North Carolina
  - Randolph Health MRI Center, Asheboro, North Carolina
  - PMG Research of Raleigh, LLC d/b/a PMG Research of Cary, Cary, North Carolina
  - Wake Radiology, Cary, North Carolina
  - Accellacare - Raleigh, Raleigh, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - Wake Radiology Diagnostic Imaging Inc, Raleigh, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Hightop Medical Research Center, Cincinnati, Ohio
  - Imaging Research Center-Cincinnati Children's, Cincinnati, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Perelman Center for Advanced Medicine, Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Clermont Radiology Orangeburg, Orangeburg, South Carolina
  - South Carolina Clinical Research LLC, Orangeburg, South Carolina
  - Tennessee Center for Clinical Trials, Tullahoma, Tennessee
  - Tullahoma HMA, LLC d\b\a Tennova HealthCare Harton, Tullahoma, Tennessee
  - Dallas Diabetes Research Center, Dallas, Texas
  - Southwest Diagnostic Imaging Center, Dallas, Texas
  - SimonMed Houston, Houston, Texas
  - Southwest Clinical Trials, Houston, Texas
  - Medical Center Hospital, Odessa, Texas
  - Permian Research Foundation, Odessa, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - National Clinical Research, Inc., Richmond, Virginia
  - Rainier Clinical Research Center, Renton, Washington
  - Bellevue Medical Imaging, Seattle, Washington
  - Universal Research Group, LLC, Tacoma, Washington
- Canada (35):
  - C-endo, Edmonton, Alberta
  - MIC Medical Imaging, Edmonton, Alberta
  - Synergy Medical Clinic, Sherwood Park, Alberta
  - Access MRI, Surrey, British Columbia
  - SMH Cardiology Clinical Trials Inc., Surrey, British Columbia
  - Nova Scotia Health Authority QE II Health Sciences Centre, Halifax, Nova Scotia
  - LMC Clinical Research Inc. (Barrie), Barrie, Ontario
  - Aggarwal and Associates Limited, Brampton, Ontario
  - LMC Clinical Research Inc. (Thornhill), Concord, Ontario
  - LMC Clinical Research Inc. (Etobicoke), Etobicoke, Ontario
  - Dawson Clinical Research, Guelph, Ontario
  - KMH Cardiology Centres Inc., Kitchener, Ontario
  - Milestone Research Inc., London, Ontario
  - Robarts Research Institute, Western University, London, Ontario
  - GNMI Medical Imaging, Mississauga, Ontario
  - GNMI MRI and CT Medical Imaging, Mississauga, Ontario
  - North York Diagnostic and Cardiac Centre, North York, Ontario
  - Bluewater Clinical Research Group Inc., Sarnia, Ontario
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario
  - Dr. Anil K. Gupta Medicine Professional Corporation, Toronto, Ontario
  - Devonshire Clinical Research Inc., Woodstock, Ontario
  - Resonance Magnetique du Saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - Ecogene-21, Chicoutimi, Quebec
  - Manna Research (Mirabel), Mirabel, Quebec
  - Recherche GCP Research, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Research Institute of the McGill University Health Center, Montreal, Quebec
  - Research Institute of the McGill University Health Centre, Montreal, Quebec
  - Radimed West Island, Pointe-Claire, Quebec
  - Diex Recherche Joliette, Saint-Charles-Borromée, Quebec
  - IRM Quebec - Complexe Synase, Québec
  - IRM Quebec Synase, Québec
  - Diex Recherche Quebec Inc., Québec
  - Centre de Recherche Saint-Louis, Québec
  - Alpha Recherche Clinique, Québec
- Poland (18):
  - NZOZ Kendron, Bialystok
  - ClinicMed Daniluk, Nowak Spolka Jawna, Bialystok
  - Malopolskie Centrum Sercowo-Naczyniowe PAKS - Chrzanow, Chrzanów
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk
  - Centrum Medyczne Enel-Med., Oddzial Alfa Plaza - Gdynia, Gdynia
  - Kardio Brynow, Katowice
  - Niepubliczny Zaklad Opieki Zdrowotnej "TERAPIA OPTIMA", Katowice
  - HELIMED Katowice - Rezonans Magnetyczny, Tomografia Komputerowa (MRI), Katowice
  - HELIMED Katowice - Rezonans Magnetyczny, Tomografia Komputerowa, Katowice
  - "TWOJA PRZYCHODNIA" Sp. z o.o., Lublin
  - Top Medical Lublin, Lublin
  - Centrum Zdrowia Metabolicznego Pawel Bogdanski, Poznan
  - Arterieart Sp. z o.o., Puszczykowo
  - SZPITAL SW. ELZBIETY W KATOWICACH Polsko-Amerykanskie Kliniki Serca, Tychy
  - Futuremeds, Wroclaw
  - Skanmex (MRI), Wroclaw
  - Wro Medica, Wroclaw
  - TOMMA Pracownia rezonansu magnetycznego we Wroclawiu, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Bergmark BA, Marston NA, Bramson CR, Curto M, Ramos V, Jevne A, Kuder JF, Park JG, Murphy SA, Verma S, Wojakowski W, Terra SG, Sabatine MS, Wiviott SD; TRANSLATE-TIMI 70 Investigators. Effect of Vupanorsen on Non-High-Density Lipoprotein Cholesterol Levels in Statin-Treated Patients With Elevated Cholesterol: TRANSLATE-TIMI 70. Circulation. 2022 May 3;145(18):1377-1386. doi: 10.1161/CIRCULATIONAHA.122.059266. Epub 2022 Apr 3. PMID 35369705
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4491011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants aged greater than equal to (>=) 40 years with dyslipidemia on a stable dose of statin (with or without ezetimibe) were included in the study. The study was conducted across 3 countries.
Pre-assignment Details: 727 participants signed the inform consent form (ICF). 391 participants were screen failures who did not meet criteria and were not enrolled. 336 participants were enrolled into the study of which 50 participants were not randomized and 286 participants were assigned to a study treatment.
Groups:
- Placebo: Participants were randomized to receive vupanorsen (PF-07285557) matched placebo subcutaneous (SC) injection. Single or double administration was given at every 2 or 4 weeks (Q2W or Q4W) to match active treatment groups. Administration locations were upper arm, thigh, or abdomen quadrant, as preferred by the participant. Treatment duration was up to 24 weeks. Participants were followed up to 12 weeks after last dose of study intervention.
- Vupanorsen: 80 mg Q4W: Participants were randomized to receive vupanorsen 80 mg single SC injection at Q4W. Administration locations were upper arm, thigh, or abdomen quadrant, as preferred by the participant. Treatment duration was up to 24 weeks. Participants were followed up to 12 weeks after last dose of study intervention.
- Vupanorsen: 60 mg Q2W: Participants were randomized to receive vupanorsen 60 mg single SC injection at Q2W. Administration locations were upper arm, thigh, or abdomen quadrant, as preferred by the participant. Treatment duration was up to 24 weeks. Participants were followed up to 12 weeks after last dose of study intervention.
- Vupanorsen: 120 mg Q4W: Participants were randomized to receive vupanorsen 60 mg double SC injection (120 mg total) in different locations at Q4W. Administration locations were upper arm, thigh, or abdomen quadrant, as preferred by the participant. Treatment duration was up to 24 weeks. Participants were followed up to 12 weeks after last dose of study intervention.
- Vupanorsen: 80 mg Q2W: Participants were randomized to receive vupanorsen 80 mg single SC injection at Q2W. Administration locations were upper arm, thigh, or abdomen quadrant, as preferred by the participant. Treatment duration was up to 24 weeks. Participants were followed up to 12 weeks after last dose of study intervention.
- Vupanorsen: 160 mg Q4W: Participants were randomized to receive vupanorsen 80 mg double SC injection (160 mg total) in different locations at Q4W. Administration locations were upper arm, thigh, or abdomen quadrant, as preferred by the participant. Treatment duration was up to 24 weeks. Participants were followed up to 12 weeks after last dose of study intervention.
- Vupanorsen: 120 mg Q2W: Participants were randomized to receive vupanorsen 60 mg double SC injection (120 mg in total) in different locations at Q2W. Administration locations were upper arm, thigh, or abdomen quadrant, as preferred by the participant. Treatment duration was up to 24 weeks. Participants were followed up to 12 weeks after last dose of study intervention.
- Vupanorsen: 160 mg Q2W: Participants were randomized to receive vupanorsen 80 mg double SC injection (160 mg in total) in different locations at Q2W. Administration locations were upper arm, thigh, or abdomen quadrant, as preferred by the participant. Treatment duration was up to 24 weeks. Participants were followed up to 12 weeks after last dose of study intervention.
Period: Treatment Period (24 Weeks)
Arm/Group | Placebo | Vupanorsen: 80 mg Q4W | Vupanorsen: 60 mg Q2W | Vupanorsen: 120 mg Q4W | Vupanorsen: 80 mg Q2W | Vupanorsen: 160 mg Q4W | Vupanorsen: 120 mg Q2W | Vupanorsen: 160 mg Q2W
Started | 44 | 23 | 24 | 23 | 45 | 45 | 46 | 36
Completed | 42 | 18 | 20 | 17 | 33 | 37 | 37 | 22
Not Completed | 2 | 5 | 4 | 6 | 12 | 8 | 9 | 14
Not completed — Other | 1 | 0 | 0 | 2 | 2 | 4 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 3 | 3 | 9 | 4 | 7 | 14
Period: Follow-up Period (12 Weeks)
Arm/Group | Placebo | Vupanorsen: 80 mg Q4W | Vupanorsen: 60 mg Q2W | Vupanorsen: 120 mg Q4W | Vupanorsen: 80 mg Q2W | Vupanorsen: 160 mg Q4W | Vupanorsen: 120 mg Q2W | Vupanorsen: 160 mg Q2W
Started | 44 (Number of participants to start this period may include participants that did not complete treatment period.) | 23 (Number of participants to start this period may include participants that did not complete treatment period.) | 24 (Number of participants to start this period may include participants that did not complete treatment period.) | 23 (Number of participants to start this period may include participants that did not complete treatment period.) | 45 (Number of participants to start this period may include participants that did not complete treatment period.) | 45 (Number of participants to start this period may include participants that did not complete treatment period.) | 46 (Number of participants to start this period may include participants that did not complete treatment period.) | 36 (Number of participants to start this period may include participants that did not complete treatment period.)
Completed | 44 | 22 | 23 | 21 | 43 | 45 | 46 | 36
Not Completed | 0 | 1 | 1 | 2 | 2 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all randomized participants.
Groups:
- Placebo: Participants were randomized to receive vupanorsen (PF-07285557) matched placebo SC injection. Single or double administration was given at every 2 or 4 weeks (Q2W or Q4W) to match active treatment groups. Administration locations were upper arm, thigh, or abdomen quadrant, as preferred by the participant. Treatment duration was up to 24 weeks. Participants were followed up to 12 weeks after last dose of study intervention.
- Total: Total of all reporting groups
Arm/Group | Placebo | Vupanorsen: 80 mg Q4W | Vupanorsen: 60 mg Q2W | Vupanorsen: 120 mg Q4W | Vupanorsen: 80 mg Q2W | Vupanorsen: 160 mg Q4W | Vupanorsen: 120 mg Q2W | Vupanorsen: 160 mg Q2W | Total
Number analyzed (Participants) | 44 | 23 | 24 | 23 | 45 | 45 | 46 | 36 | 286
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.23 (8.09) | 65.78 (7.27) | 64.21 (9.92) | 61.04 (9.31) | 63.38 (8.41) | 63.09 (8.80) | 62.74 (8.64) | 64.47 (7.74) | 63.57 (8.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 7 | 9 | 24 | 17 | 20 | 19 | 126
  Male | 27 | 10 | 17 | 14 | 21 | 28 | 26 | 17 | 160
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 1 | 6 | 4 | 6 | 2 | 1 | 27
  Not Hispanic or Latino | 39 | 21 | 23 | 17 | 41 | 39 | 44 | 35 | 259
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 2 | 2 | 1 | 3 | 0 | 4 | 4 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 4 | 1 | 4 | 1 | 12
  White | 38 | 20 | 21 | 21 | 38 | 44 | 37 | 31 | 250
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Non-High-Density Lipoprotein-Cholesterol (Non-HDL-C) at Week 24
Description: Fasting was required at least 10 hours before blood sample collection. Baseline was calculated using the average of all values obtained at Screening and on Day 1 prior to dosing.
Time Frame: Baseline, Week 24
Population: Full analysis set primary (FAS_primary) included all participants randomized to study intervention and who took at least 1 dose of study intervention, had a baseline measurement and at least one post-baseline measurement with all observations that occurred after discontinuation of treatment or after initiation of severe hypertriglyceridemia excluded.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Vupanorsen: 80 mg Q4W | Vupanorsen: 60 mg Q2W | Vupanorsen: 120 mg Q4W | Vupanorsen: 80 mg Q2W | Vupanorsen: 160 mg Q4W | Vupanorsen: 120 mg Q2W | Vupanorsen: 160 mg Q2W
Number analyzed (Participants) | 44 | 23 | 23 | 23 | 42 | 45 | 46 | 35
Percent change | -1.1 (2.76) | -23.5 (4.08) | -23.2 (4.02) | -25.3 (4.23) | -28.8 (3.02) | -27.8 (2.88) | -25.8 (2.84) | -27.6 (3.57)
Statistical Analysis 1: Comparison: Placebo vs Vupanorsen: 80 mg Q4W; Test type: Other; p < 0.001, Mixed Models Analysis; MMRM with baseline value, treatment, visit, interaction term of treatment by visit as fixed effects and unstructured covariance structure was used; Least Square (LS) Mean difference = -22.4, 95% CI 2-sided [-32.1 to -12.7], Standard Error of Mean 4.93
Statistical Analysis 2: Comparison: Placebo vs Vupanorsen: 60 mg Q2W; Test type: Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -22.0, 95% CI 2-sided [-31.7 to -12.4], Standard Error of Mean 4.88
Statistical Analysis 3: Comparison: Placebo vs Vupanorsen: 120 mg Q4W; Test type: Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -24.1, 95% CI 2-sided [-34.1 to -14.2], Standard Error of Mean 5.05
Statistical Analysis 4: Comparison: Placebo vs Vupanorsen: 80 mg Q2W; Test type: Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -27.7, 95% CI 2-sided [-35.7 to -19.6], Standard Error of Mean 4.09
Statistical Analysis 5: Comparison: Placebo vs Vupanorsen: 160 mg Q4W; Test type: Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -26.6, 95% CI 2-sided [-34.5 to -18.8], Standard Error of Mean 3.98
Statistical Analysis 6: Comparison: Placebo vs Vupanorsen: 120 mg Q2W; Test type: Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -24.7, 95% CI 2-sided [-32.5 to -16.9], Standard Error of Mean 3.96
Statistical Analysis 7: Comparison: Placebo vs Vupanorsen: 160 mg Q2W; Test type: Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -26.5, 95% CI 2-sided [-35.4 to -17.6], Standard Error of Mean 4.51

2. Secondary Outcome: Percent Change From Baseline in Triglyceride (TG), Apolipoprotein B (ApoB), Low-Density Lipoprotein-Cholesterol (LDL-C), and Non-HDL-C at Week 16
Description: Blood samples were collected from participants in a fasted state for the measurement of TG, ApoB, HDL-C and LDL-C. Fasting was required at least 10 hours before blood sample collection. Non-HDL-C was calculated as total cholesterol minus HDL cholesterol. Baseline was calculated using the average of all values obtained at Screening and on Day 1 prior to dosing.
Time Frame: Baseline, Week 16
Population: FAS included all participants randomized to study intervention and who took at least 1 dose of study intervention and had a baseline measurement and at least one post-baseline measurement. Here, "Number Analyzed" signifies participants evaluable for specific rows.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Vupanorsen: 80 mg Q4W | Vupanorsen: 60 mg Q2W | Vupanorsen: 120 mg Q4W | Vupanorsen: 80 mg Q2W | Vupanorsen: 160 mg Q4W | Vupanorsen: 120 mg Q2W | Vupanorsen: 160 mg Q2W
Number analyzed (Participants) | 44 | 23 | 24 | 23 | 43 | 45 | 46 | 36
Percent change
  TG: number analyzed (Participants) | 43 | 22 | 23 | 21 | 40 | 43 | 44 | 35
  TG | -2.53 (31.247) | -42.17 (28.081) | -44.71 (22.725) | -39.57 (32.546) | -49.21 (21.049) | -40.33 (21.311) | -50.55 (20.234) | -55.76 (14.625)
  ApoB: number analyzed (Participants) | 41 | 21 | 22 | 22 | 40 | 44 | 43 | 34
  ApoB | 0.66 (20.372) | -12.12 (15.839) | -12.30 (12.604) | -10.41 (17.067) | -10.40 (14.690) | -10.42 (19.332) | -11.74 (15.560) | -6.76 (18.890)
  LDL-C: number analyzed (Participants) | 41 | 22 | 22 | 20 | 40 | 42 | 44 | 35
  LDL-C | -1.42 (24.092) | -10.40 (31.199) | -12.61 (21.904) | -2.09 (26.921) | -11.38 (22.001) | -10.88 (26.640) | -13.78 (19.861) | -6.30 (29.825)
  Non-HDL-C: number analyzed (Participants) | 43 | 22 | 23 | 21 | 40 | 43 | 44 | 35
  Non-HDL-C | -3.25 (21.631) | -21.65 (24.347) | -24.71 (16.678) | -20.06 (16.698) | -24.79 (18.266) | -21.68 (23.898) | -27.23 (12.799) | -22.44 (24.145)

3. Secondary Outcome: Percent Change From Baseline in TG, ApoB, and LDL-C at Week 24
Description: Fasting was required for all lipid measures at least 10 hours before blood sample collection. Baseline was calculated using the average of all values obtained at Screening and on Day 1 prior to dosing.
Time Frame: Baseline, Week 24
Population: FAS_primary included all participants randomized to study intervention and who took at least 1 dose of study intervention, had a baseline measurement and at least one post-baseline measurement with all observations that occurred after discontinuation of treatment or after initiation of severe hypertriglyceridemia excluded. Here, "Number Analyzed" signifies participants evaluable for specific rows.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Vupanorsen: 80 mg Q4W | Vupanorsen: 60 mg Q2W | Vupanorsen: 120 mg Q4W | Vupanorsen: 80 mg Q2W | Vupanorsen: 160 mg Q4W | Vupanorsen: 120 mg Q2W | Vupanorsen: 160 mg Q2W
Number analyzed (Participants) | 44 | 23 | 23 | 23 | 42 | 45 | 46 | 35
Percent change
  TG | -1.8 (3.71) | -45.8 (5.53) | -45.6 (5.50) | -43.1 (5.76) | -52.3 (4.10) | -47.7 (3.90) | -52.5 (3.85) | -58.6 (4.90)
  ApoB: number analyzed (Participants) | 42 | 22 | 22 | 23 | 41 | 45 | 44 | 35
  ApoB | 0.3 (2.46) | -14.8 (3.60) | -10.3 (3.57) | -11.2 (3.76) | -12.2 (2.68) | -12.2 (2.55) | -5.6 (2.57) | -8.1 (3.17)
  LDL-C: number analyzed (Participants) | 43 | 23 | 22 | 22 | 42 | 43 | 46 | 35
  LDL-C | -1.2 (3.69) | -11.2 (5.41) | -9.1 (5.52) | -12.7 (5.63) | -17.3 (4.00) | -15.7 (3.92) | -9.1 (3.77) | -10.2 (4.74)
Statistical Analysis 1: Comparison: Placebo vs Vupanorsen: 80 mg Q4W; TG; Test type: Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -44.0, 95% CI 2-sided [-57.1 to -30.8], Standard Error of Mean 6.66
Statistical Analysis 2: Comparison: Placebo vs Vupanorsen: 60 mg Q2W; TG; Test type: Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -43.8, 95% CI 2-sided [-56.9 to -30.7], Standard Error of Mean 6.64
Statistical Analysis 3: Comparison: Placebo vs Vupanorsen: 120 mg Q4W; TG; Test type: Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -41.3, 95% CI 2-sided [-54.8 to -27.8], Standard Error of Mean 6.85
Statistical Analysis 4: Comparison: Placebo vs Vupanorsen: 80 mg Q2W; TG; Test type: Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -50.5, 95% CI 2-sided [-61.4 to -39.6], Standard Error of Mean 5.54
Statistical Analysis 5: Comparison: Placebo vs Vupanorsen: 160 mg Q4W; TG; Test type: Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -45.9, 95% CI 2-sided [-56.5 to -35.2], Standard Error of Mean 5.38
Statistical Analysis 6: Comparison: Placebo vs Vupanorsen: 120 mg Q2W; TG; Test type: Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -50.7, 95% CI 2-sided [-61.2 to -40.1], Standard Error of Mean 5.35
Statistical Analysis 7: Comparison: Placebo vs Vupanorsen: 160 mg Q2W; TG; Test type: Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -56.8, 95% CI 2-sided [-68.9 to -44.7], Standard Error of Mean 6.14
Statistical Analysis 8: Comparison: Placebo vs Vupanorsen: 80 mg Q4W; ApoB; Test type: Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -15.1, 95% CI 2-sided [-23.7 to -6.5], Standard Error of Mean 4.36
Statistical Analysis 9: Comparison: Placebo vs Vupanorsen: 60 mg Q2W; ApoB; Test type: Other; p = 0.015, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -10.6, 95% CI 2-sided [-19.2 to -2.1], Standard Error of Mean 4.34
Statistical Analysis 10: Comparison: Placebo vs Vupanorsen: 120 mg Q4W; ApoB; Test type: Other; p = 0.011, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -11.5, 95% CI 2-sided [-20.3 to -2.7], Standard Error of Mean 4.49
Statistical Analysis 11: Comparison: Placebo vs Vupanorsen: 80 mg Q2W; ApoB; Test type: Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -12.5, 95% CI 2-sided [-19.7 to -5.3], Standard Error of Mean 3.64
Statistical Analysis 12: Comparison: Placebo vs Vupanorsen: 160 mg Q4W; ApoB; Test type: Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -12.6, 95% CI 2-sided [-19.5 to -5.6], Standard Error of Mean 3.54
Statistical Analysis 13: Comparison: Placebo vs Vupanorsen: 120 mg Q2W; ApoB; Test type: Other; p = 0.095, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -6.0, 95% CI 2-sided [-13.0 to 1.0], Standard Error of Mean 3.56
Statistical Analysis 14: Comparison: Placebo vs Vupanorsen: 160 mg Q2W; ApoB; Test type: Other; p = 0.036, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -8.5, 95% CI 2-sided [-16.4 to -0.6], Standard Error of Mean 4.01
Statistical Analysis 15: Comparison: Placebo vs Vupanorsen: 80 mg Q4W; LDL-C; Test type: Other; p = 0.129, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -10.0, 95% CI 2-sided [-22.9 to 2.9], Standard Error of Mean 6.55
Statistical Analysis 16: Comparison: Placebo vs Vupanorsen: 60 mg Q2W; LDL-C; Test type: Other; p = 0.238, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -7.9, 95% CI 2-sided [-21.0 to 5.2], Standard Error of Mean 6.65
Statistical Analysis 17: Comparison: Placebo vs Vupanorsen: 120 mg Q4W; LDL-C; Test type: Other; p = 0.090, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -11.4, 95% CI 2-sided [-24.7 to 1.8], Standard Error of Mean 6.73
Statistical Analysis 18: Comparison: Placebo vs Vupanorsen: 80 mg Q2W; LDL-C; Test type: Other; p = 0.004, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -16.0, 95% CI 2-sided [-26.7 to -5.3], Standard Error of Mean 5.44
Statistical Analysis 19: Comparison: Placebo vs Vupanorsen: 160 mg Q4W; LDL-C; Test type: Other; p = 0.008, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -14.5, 95% CI 2-sided [-25.1 to -3.9], Standard Error of Mean 5.38
Statistical Analysis 20: Comparison: Placebo vs Vupanorsen: 120 mg Q2W; LDL-C; Test type: Other; p = 0.136, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -7.9, 95% CI 2-sided [-18.3 to 2.5], Standard Error of Mean 5.28
Statistical Analysis 21: Comparison: Placebo vs Vupanorsen: 160 mg Q2W; LDL-C; Test type: Other; p = 0.138, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -9.0, 95% CI 2-sided [-20.8 to 2.9], Standard Error of Mean 6.01

4. Secondary Outcome: Percent Change From Baseline in Angiopoietin-like Protein 3 (ANGPTL3) at Week 16
Description: ANGPTL3 is a protein primarily synthesized and secreted by the liver and is a member of the angiopoietin-like family of proteins. Blood samples were collected from participants in a fasted state for the measurement of ANGPTL3. Fasting was required at least 10 hours before blood sample collection. Baseline was calculated using the average of all values obtained at Screening and on Day 1 prior to dosing.
Time Frame: Baseline, Week 16
Population: FAS included all participants randomized to study intervention and who took at least 1 dose of study intervention and had a baseline measurement and at least one post-baseline measurement. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Vupanorsen: 80 mg Q4W | Vupanorsen: 60 mg Q2W | Vupanorsen: 120 mg Q4W | Vupanorsen: 80 mg Q2W | Vupanorsen: 160 mg Q4W | Vupanorsen: 120 mg Q2W | Vupanorsen: 160 mg Q2W
Number analyzed (Participants) | 41 | 21 | 21 | 21 | 39 | 44 | 41 | 32
Percent change | 9.14 (36.729) | -51.12 (30.444) | -63.61 (16.934) | -58.19 (22.175) | -65.56 (21.908) | -60.35 (21.040) | -77.55 (15.469) | -75.14 (23.549)

5. Secondary Outcome: Percent Change From Baseline in ANGPTL3 at Week 24
Description: as for outcome 4
Time Frame: Baseline, Week 24
Population: FAS_primary included all participants randomized to study intervention and who took at least 1 dose of study intervention, had a baseline measurement and at least one post-baseline measurement with all observations that occurred after discontinuation of treatment or after initiation of severe hypertriglyceridemia excluded. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Vupanorsen: 80 mg Q4W | Vupanorsen: 60 mg Q2W | Vupanorsen: 120 mg Q4W | Vupanorsen: 80 mg Q2W | Vupanorsen: 160 mg Q4W | Vupanorsen: 120 mg Q2W | Vupanorsen: 160 mg Q2W
Number analyzed (Participants) | 42 | 22 | 21 | 22 | 40 | 45 | 42 | 33
Percent change | 13.3 (3.36) | -56.6 (4.92) | -66.3 (5.01) | -63.8 (5.22) | -73.0 (3.76) | -67.1 (3.46) | -78.9 (3.58) | -81.9 (4.48)
Statistical Analysis 1: Comparison: Placebo vs Vupanorsen: 80 mg Q4W; Test type: Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -69.9, 95% CI 2-sided [-81.6 to -58.1], Standard Error of Mean 5.97
Statistical Analysis 2: Comparison: Placebo vs Vupanorsen: 60 mg Q2W; Test type: Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -79.6, 95% CI 2-sided [-91.5 to -67.7], Standard Error of Mean 6.03
Statistical Analysis 3: Comparison: Placebo vs Vupanorsen: 120 mg Q4W; Test type: Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -77.1, 95% CI 2-sided [-89.4 to -64.9], Standard Error of Mean 6.22
Statistical Analysis 4: Comparison: Placebo vs Vupanorsen: 80 mg Q2W; Test type: Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -86.3, 95% CI 2-sided [-96.2 to -76.3], Standard Error of Mean 5.04
Statistical Analysis 5: Comparison: Placebo vs Vupanorsen: 160 mg Q4W; Test type: Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -80.4, 95% CI 2-sided [-89.9 to -70.9], Standard Error of Mean 4.82
Statistical Analysis 6: Comparison: Placebo vs Vupanorsen: 120 mg Q2W; Test type: Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -92.2, 95% CI 2-sided [-101.9 to -82.6], Standard Error of Mean 4.92
Statistical Analysis 7: Comparison: Placebo vs Vupanorsen: 160 mg Q2W; Test type: Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean difference = -95.2, 95% CI 2-sided [-106.2 to -84.2], Standard Error of Mean 5.59

ADVERSE EVENTS:
Time Frame: From start of study intervention up to 12 weeks after last dose of study intervention (maximum for 36 weeks)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Placebo | Vupanorsen: 80 mg Q4W | Vupanorsen: 60 mg Q2W | Vupanorsen: 120 mg Q4W | Vupanorsen: 80 mg Q2W | Vupanorsen: 160 mg Q4W | Vupanorsen: 120 mg Q2W | Vupanorsen: 160 mg Q2W
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/23 | 0/24 | 0/23 | 0/45 | 0/45 | 0/46 | 0/36
Serious Adverse Events (participants affected / at risk) | 4/44 | 2/23 | 2/24 | 0/23 | 6/45 | 1/45 | 3/46 | 1/36
Other Adverse Events (participants affected / at risk) | 31/44 | 15/23 | 17/24 | 12/23 | 30/45 | 28/45 | 29/46 | 31/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=44) | Vupanorsen: 80 mg Q4W (N=23) | Vupanorsen: 60 mg Q2W (N=24) | Vupanorsen: 120 mg Q4W (N=23) | Vupanorsen: 80 mg Q2W (N=45) | Vupanorsen: 160 mg Q4W (N=45) | Vupanorsen: 120 mg Q2W (N=46) | Vupanorsen: 160 mg Q2W (N=36)
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=44) | Vupanorsen: 80 mg Q4W (N=23) | Vupanorsen: 60 mg Q2W (N=24) | Vupanorsen: 120 mg Q4W (N=23) | Vupanorsen: 80 mg Q2W (N=45) | Vupanorsen: 160 mg Q4W (N=45) | Vupanorsen: 120 mg Q2W (N=46) | Vupanorsen: 160 mg Q2W (N=36)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Brugada syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myocardial injury (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ulcerative keratitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acid peptic disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dental necrosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 1 | 1 | 2 | 2
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 2 | 1 | 0 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 1 | 0 | 1 | 2 | 3 | 0
Hunger (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Injection site dermatitis (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Injection site erythema (General disorders) | 0 | 1 | 1 | 2 | 2 | 1 | 3 | 4
Injection site pain (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Injection site rash (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 1 | 3 | 4 | 4 | 4 | 6 | 8
Injection site recall reaction (General disorders) | 0 | 0 | 2 | 1 | 2 | 0 | 5 | 3
Injection site vesicles (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Therapeutic response unexpected (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nonalcoholic fatty liver disease (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infection parasitic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 1 | 1 | 1 | 3 | 1 | 1 | 3
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 0 | 1 | 1 | 4 | 9
Albumin urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 4
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood potassium abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Creatinine renal clearance abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QRS complex prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematocrit increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 3
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Magnetic resonance imaging spinal abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mean cell haemoglobin concentration decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mean cell volume increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urine albumin/creatinine ratio abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine albumin/creatinine ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urine analysis abnormal (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 6
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 4 | 1 | 3 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 3 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 0 | 3 | 0 | 2 | 0
Plantar fascial fibromatosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0 | 6 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 1 | 1 | 2 | 3 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Adjustment disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Microalbuminuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urge incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Genital atrophy (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT04516291/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/91/NCT04516291/SAP_001.pdf